CLINICAL TRIAL: NCT03541278
Title: A Prospective Multicenter Clinical Trial of Internal Mammary Sentinel Lymph Node Biopsy With Modified Injection Technique for Early Breast Cancer
Brief Title: Internal Mammary Sentinel Lymph Node Biopsy With Modified Injection Technique
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Recruiting
Sponsor: Shandong Cancer Hospital and Institute (Other)
Collaborators: The Affiliated Hospital of Qingdao University (Other); Henan Cancer Hospital (Other Government)
Responsible Party: Principal Investigator, Yongsheng Wang, Director, Head of Breast Cancer Center, Principal Investigator, Clinical Professor, Shandong Cancer Hospital and Institute
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Diagnostic
Other Study IDs: PMCT-IMSLNB-MIT
Record Dates: First submitted 2018-05-18; First posted 2018-05-30 (Actual); Last update posted 2018-05-30 (Actual); Status verified 2018-05

CONDITIONS: Breast Cancer
Keywords: Breast Cancer; Internal Mammary Lymph Node; Internal Mammary Sentinel Lymph Node Biopsy; Detection Rate
MeSH Terms: conditions — Breast Neoplasms

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (1):
- IM-SLNB with MIT (Experimental): The radiotracer was injected with our modified injection technique (MIT) (periareolar intraparenchymal, high volume and ultrasonographic guidance). Internal mammary sentinel lymph node biopsy (IM-SLNB) was performed for patients with internal mammary visualized.
  Interventions: Procedure: MIT; Procedure: IM-SLNB

INTERVENTIONS:
Procedure: MIT — periareolar intraparenchymal, high volume and ultrasonographic guidance
  Other Names: Modified Injection Technique
Procedure: IM-SLNB — IM-SLNB was performed for IMLN visualized patients
  Other Names: Internal Mammary Sentinel Lymph Node Biopsy

SUMMARY:
Internal Mammary Lymph Node (IMLN) and Axillary Lymph Node (ALN) are regarded as "the first station" of lymphatic drainage in breast cancer, serving as an important reference for lymph staging and decision-making. Although the concept of Internal Mammary Sentinel Lymph Node Biopsy (IM-SLNB) has been included in the AJCC guidelines since the 6th edition, technical bottlenecks and clinical benefits still remained to be the main reasons limiting its clinical application:

Technical bottlenecks: In previous clinical practice, the internal mammary visualization rate was very low (13% on average, 0% -37%) under the guidance of the traditional radionuclide injection technique, which became a technology bottleneck restricting the widespread of IM-SLNB. After continuous exploration, our center invented the "modified injection technique" of injecting the nuclide tracer into the mammary gland layer at 6 and 12 o'clock around the areolar under the guidance of ultrasound, as well as increasing the injection volume to increase the local tension. A high internal mammary imaging rate of 71% was obtained, which laid a foundation for the further study and clinical application of IM-SLNB.

Clinical benefits: The IM-SLNB is a method to assess IMLN metastatic status in a minimally invasive way, which may improve the system of regional staging and guide precise IMLN treatment. However, based on the current IM-SLNB indication, the internal mammary metastasis rate was only 8%-15%, and it only had little influence on treatment strategy, which led to the controversy of its clinical application. Previous studies of extended radical mastectomy showed that in ALN positive patients the IMLN metastasis rate was 28-52%, while in ALN negative patients the metastasis rate was only 5-17%. Therefore, the continuation of the previous A-SLNB indication (clinical ALN negative) to IM-SLNB is apparently not in line with the current clinical practice, but further evaluation of internal mammary metastasis status in clinical ALN positive patients may receive greater benefit.

This prospective multicenter study attempted to perform IM-SLNB with our modified injection technique both in clinical ALN negative and positive patients for the first time. Through analyzing metastasis rate of IMLN as well as the influences it had on decision making, we hoped to develop more accurate indication for IM-SLNB and guide the individualized precise treatment of IMLN.

DETAILED DESCRIPTION:
Tracer injection and Lymphatic imaging: The radionuclide tracer (99mTc-Sulfur colloid) was prepared by the Nuclear Medicine Department and the sulfur colloid kit (equipped with a filter of 220 nm in diameter to control the size of colloidal particles) was prepared by Beijing Xinkesida company. All patients were injected with 99mTc-Sulfur colloid (1.0~1.2ml/29.6~55.5MBq) in periareolar parenchyma gland under the guidance of ultrasound using the "new injection technique" 3-18h before surgery. SPECT / CT lymphoscintigraphy was performed 30 min before surgery, and the radioactive concentration ("hot spot") near the sternum was defined as IMSLN positive.

IM-SLNB: After modified radical mastectomy / breast-conserving radical surgery, intraoperative γ-detector (Neoprobe 2000, Johnson& Johnson Company) was used to locate IM-SLN, and intercostal IM-SLNB was performed: open pectoralis major muscle, expose the parasternal intercostal space at the corresponding intercostal level (if the patient underwent breast-conserving surgery and the tumor was located in the lateral quadrant, an additional 3 cm of skin incision was required), cut the intercostal muscle at radioactive concentration site parallel to the rib, search and locate IMSLN with gamma detector, dissect precisely to avoid injury of internal mammary arteries and veins, and then sent the removed tissue to routine pathological examination.

Pathologic diagnosis: IMSLN was divided into 2mm tissue fragments according to the long axis (short diameter < 2 mm, no division), every tissue fragment required one layer of routine HE staining pathological examination. In this study, metastasis > 0.2mm was defined as IMSLN positive, while solitary tumor cell was defined as IMSLN negative. Further IHC detection of CK-9 was required if the IMSLN was HE staining negative to exclude micrometastasis.

ELIGIBILITY:
Inclusion Criteria:

* Patients with preoperative pathology confirmed invasive breast cancer;
* Clinical T1-3 N0-3 M0 (with positive fine-needle aspiration result in their clinical or ultrasonic suspicious axillary lymph node ; no clinical or radiologic evidence of distant metastases);
* Be able and willing to sign informed consent forms.

Exclusion Criteria:

* Patients with enlarged internal mammary nodes by imaging;
* Patients who have received neoadjuvant therapy (including neoadjuvant chemotherapy and / or endocrine therapy);
* Patients with a previous history of breast cancer (recurrence of breast cancer and contralateral breast cancer);
* Patients with a history of other malignancies;
* Patients who have had previous surgery in axillary or internal mammary;
* Patients in pregnancy and lactation;
* Patients participant in other clinical trials that will have an impact on the results of this study.

Ages: 18 Years to 70 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 350 (Estimated)
Dates: Start 2018-07-01 (Estimated); Primary Completion 2020-06-30 (Estimated); Study Completion 2020-12-31 (Estimated)

PRIMARY OUTCOMES:
Visualization Rate | 2 year
  The internal mammary sentinel lymph node visualization rate with our modified injection techniques

SECONDARY OUTCOMES:
Success rate of IM-SLNB | 2 year
  Success rate of IM-SLNB in the IMSLN visualization patients who receive IM-SLNB
Frequency and Severity of Complications with IM-SLNB | 2 year
  IM-SLNB complications in the patients who receive IM-SLNB
Metastasis Rate of IMSLN | 2 year
  Metastasis rate of IMSLN in clinically axillary node-negative and clinically axillary node-positive patients
Clinical Benefits | 2 year
  staging and treatment change rate

CONTACTS AND LOCATIONS:
Overall Officials: Yong-Sheng Yong-Sheng, MD, Study Chair — Shandong Cancer Hospital and Institute
Locations (1):
- Shandong Cancer Hospital and Institute, Jinan, Shandong, China

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Qiu PF, Liu JJ, Liu YB, Yang GR, Sun X, Wang YS. A modified technology could significantly improve the visualization rate of the internal mammary sentinel lymph nodes in breast cancer patients. Breast Cancer Res Treat. 2012 Nov;136(1):319-21. doi: 10.1007/s10549-012-2203-5. Epub 2012 Sep 6. No abstract available. PMID 22956005